CLINICAL TRIAL: NCT00311233
Title: Recurrent Abdominal Pain in Childhood, Characteristics and Course
Brief Title: Recurrent Abdominal Pain in Childhood -Characteristics and Course
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Regionsenter for barn og unges psykiske helse (Other)
Other Study IDs: 150063
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Abdominal Pain
Keywords: child; psychosocial; predictors; cohort; recurrent
MeSH Terms: conditions — Abdominal Pain; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All patients have blood tests for hemoglobin, total leucocyte and differential count, sedimention rate, C-reactive protein, total IgE and IgE screen for food allergies, and antiendomysial and antigliadin antibodies (IgG and IgA) and anti-tissue transglutaminase antibodies for celiac disease. Furthermore, urine analyses for protein, blood and and leucocytes, three stool specimen for occult blood and one stool specimen for quantification of calprotectin.

SUMMARY:
Recurrent abdominal pain (RAP) is a common complaint in childhood. Identification of the processes that maintain illness is important.

The purpose of this study is to get more knowledge about characteristics of children with recurrent abdominal pain and their parents, and about the course of their pain. These results may be important to identify children who need treatment.

DETAILED DESCRIPTION:
BACKGROUND:

Recurrent abdominal pain (RAP), mainly constituted by functional gastrointestinal disorders (FGID), affects a significant number of children, and is a result of a complex interaction between biopsychosocial factors. Despite the seemingly benign nature of RAP, in some children RAP is associated with school absenteeism, functional impairment and frequent doctor visits. Identification of the processes that maintain illness is important. These results may be important to identify children who need treatment.

AIMS:

The aims of this study are to characterize children with RAP (in four out-patient clinics) and their parents, describe outcome and determine predictors of persistent RAP in children.

SAMPLE:

150 pediatric patients (4-15 years), their parents and teachers. Consecutive new patients referred to four pediatric out-patients clinics for evaluation of abdominal pain (primary complaint). Patients with RAP (abdominal pain at least once a month, in three consecutive months during the last year, and whose pains are severe enough to affect daily activity) are eligible.

DESIGN: A prospective cohort study.

MEASUREMENT:

All pediatric patients will undergo a complete physical examination emphasizing diagnosing organic illness and FGID according to the international ROME classification. Routine laboratory will be done. A protocol to identify somatic causes is part of the study. In addition, parents will complete validated questionnaires regarding their child's physical/psychological health, temperamental characteristics and social skills and also psychosocial conditions concerning them selves. Self-report regarding the same aspects will be obtained from children above 8-9 years.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive new pediatric patients (4-15 years) referred by their general practitioners to four pediatric out-patient clinics in Innlandet Hospital Health Authorities for evaluation of recurrent abdominal pain.

Exclusion Criteria:

* Known organic diagnosis for abdominal pain
* Language problems (which will interfere completing questionnaires)

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Consecutive new pediatric patients (4-15 years) referred by their general practitioners to four pediatric out-patient clinics in Innlandet Hospital Health Authorities for evaluation of recurrent abdominal pain.
Enrollment: 152 (Actual)
Dates: Start 2006-02; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trond Markestad, MD, Phd, Study Chair — Eastern Norway Health Authorities, Innlandet Hospital Health Authorities
Locations (1):
- Division of women and child and Division of Child and Adolescent Psychiatry, Innlandet Hospital Health Authorities, Gjøvik, Norway